CLINICAL TRIAL: NCT05640986
Title: Use of BART Coupled With EEG in the Early Diagnosis of Behavioral Disorders in Parkinson's Disease: a Pilot Study
Brief Title: Use of BART Coupled With EEG in the Early Diagnosis of Behavioral Disorders in Parkinson's Disease
Acronym: COMPARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021/615
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Risky behaviors assessed through BART-EEG among Parkinsonian patients newly treated with dopaminergic agonists
  Interventions: Behavioral: BART-EEG at V1 + V2
- Control (Active Comparator): Risky behaviors assessed through BART-EEG among healthy volunteers
  Interventions: Behavioral: BART-EEG at V1 only

INTERVENTIONS:
Behavioral: BART-EEG at V1 + V2 — Balloon Analogue Risk Task coupled to Electroencephalogram (BART-EEG) at V1 + V2 for Parkinsonian patients
  Arms: Patients
Behavioral: BART-EEG at V1 only — Balloon Analogue Risk Task coupled to Electroencephalogram (BART-EEG) at V1 only for healthy volunteers
  Arms: Control

SUMMARY:
The Balloon Analogue Risk Task [BART] is an experimental task modelizing risky behaviors. In Parkinson disease, the correlation between BART and modifications of cerebral activity in ventral striatum has been shown. BART thus seems to be particularly adapted for modelization of HYPERdopaminergic behavioral disorders [TYPER] into Parkinsonian patients. Previously, a version of the BART performed with EEG has been specifically developped by the Centre d'Investigation Clinique of Besançon University Hospital, in collaboration with the Clinical and integrative neurosciences laboratory. Preliminary data suggest that the analysis of evoked potentials including Feedback-related Negativity [FRN], P300 wave, and Reward Positivity [RewP], could help assessing the motivational and attentional attributes of decision making and the delayed treatment of any reward.

The hypothesis of the study that the EEG version of the BART could help predicting the risk to develop TYPER into Parkinsonian patients treated by dopaminergic in routine care.

ELIGIBILITY:
Inclusion Criteria:

* Probable Diagnosis of Parkinson's disease according to the Movement Disorder Society criteria
* Parkinson disease appeared ≤ 60 years old
* Disease evolving since ≥ 5 years
* Daily dose for du dopaminergic treatment ≥ 200mg/day DOPA equivalent
* Patients requiring in routine care the introduction or increase of dopaminergic agonists treatment because of:

  1. HYPOdopaminergic behavioral syndrome [TYPO] including apathy, anxiety, depression and/or
  2. motor syndrome insufficiently controlled by dopaminergic treatment (akinesia, rigidity, tremor)

Exclusion Criteria:

* Cognitive disorders (Montreal Cognitive Assessment [MoCA] < 25/30)
* Parkinson disease psychosis
* HYPERdopaminergic behavioral disorders [TYPER] defined by a score ≥ 2 at at least 1 item of HYPERdopaminergic behavioral spectrum of Parkinson disease
* Contraindications for dopaminergic agonists
* Patient treated with deep brain stimulation
* Serious psychiatric comorbidity (major depressive episode according to Diagnostic and Statistical Manual of Mental Disorders [DSM] V criteria, suicidal patient, other active psychosis, etc.)
* Unstabilized psychotropic treatment
* Pregnant or breastfeeding women

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Area under curve for dopaminergic agonist treatment | Month 9
  Area Under the Curve / Receiver Operating Characteristic Curve [AUC-ROC] of [FRN] amplitude measured at baseline for TYPER risk 9 months after introduction or increase of dopaminergic agonist treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu BEREAU, MD, Principal Investigator — CHU de Besançon